CLINICAL TRIAL: NCT04497090
Title: Non-invasive Ventilation With Automatic Expiratory Positive Airway Pressure Titration to Abolish Tidal Expiratory Flow Limitation in COPD Patients With Chronic Hypercapnia
Brief Title: Adaptive Non-invasive Ventilation to Abolish Tidal Flow Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Politecnico di Milano (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Raffaele Dellaca, Prof, Politecnico di Milano
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Polimi
Record Dates: First submitted 2020-07-25; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hypercapnia; Ventilator Lung
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-EPAP (Active Comparator): EPAP was kept fixed at the prescribed level throughout the night
  Interventions: Device: fixed-EPAP
- Auto-EPAP (Experimental): EPAP was continuously adjusted using the experimental approach aimed at abolishing tidal expiratory flow limitation
  Interventions: Device: auto-EPAP

INTERVENTIONS:
Device: fixed-EPAP — In the fixed-EPAP mode, the device kept EPAP fixed at the prescribed value
  Arms: Fixed-EPAP
Device: auto-EPAP — In the Auto-EPAP mode, the device automatically adjusted EPAP to the minimum level able to abolish tidal expiratory flow limitation.
  Arms: Auto-EPAP

SUMMARY:
This study aimed to evaluate the effects of a novel automatic non-invasive ventilation (NIV) mode that continuously adjusts expiratory positive airway pressure (EPAP) to the lowest value that abolishes tidal expiratory flow limitation. The investigators conducted a prospective, randomized, cross-over study on stable chronic obstructive pulmonary disease (COPD) patients. Patients were studied in the hospital during two non-consecutive nights while using either fixed or adaptive EPAP. The primary outcome was the transcutaneous partial pressure of carbon dioxide. Secondary outcomes were: oxygen saturation, breathing pattern, oscillatory mechanics, patient-ventilation asynchronies, sleep quality and sleep-related respiratory events.

DETAILED DESCRIPTION:
Study design: prospective, randomized, cross-over study. Study population: moderate to severe COPD patients, long-term users of nocturnal non-invasive ventilation for chronic hypercapnic respiratory failure. Inclusion criteria: age<85 years; presence of tidal expiratory flow limitation in the supine position at an expiratory positive airway pressure of 4 cmH2O. Exclusion criteria: COPD exacerbation within the past two months; acute illness; clinical instability.

Study protocol: Patients were studied in the hospital over 2 non-consecutive nights while using either fixed or automatic EPAP.

Ventilation strategy: pressure-controlled NIV was delivered using a non-commercial version of BiPAP Synchrony Ventilator (Philips-Respironics) via an unvented facial mask (AMARA, Philips-Respironics). The ventilator evaluated the presence of tidal expiratory flow limitation by the forced oscillation technique. In the automatic-EPAP mode, the ventilator continuously adjusted EPAP to the minimum level able to abolish tidal expiratory flow limitation, with a minimum EPAP of 4 cmH2O and keeping the pressure support constant.

Measurements: During each study night, the investigators recorded transcutaneous partial pressure of carbon dioxide and oxygen saturation (TOSCA, Radiometer) continuously. Airway opening pressure, flow and volume tracings were exported from the ventilator. Full laboratory polysomnography (Alice5, Philips-Respironics) was performed according to the American Academy of Sleep Medicine recommendations.

Data analysis: the investigators compared parameters from the two nights using Wilcoxon signed-rank test. P-values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe COPD (GOLD 2017);
* long-term users of nocturnal non-invasive ventilation for chronic hypercapnic respiratory failure;
* presence of tidal expiratory flow limitation in the supine position at an expiratory positive airway pressure of 4 cmH2O.

Exclusion Criteria:

* COPD exacerbation within the past two months;
* acute illness;
* clinical instability.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Mean transcutaneous partial pressure of carbon dioxide (PtcCO2) | Overnight (about 8 hours)
  The partial pressure of carbon dioxide measures the efficacy of ventilation. Reducing PCO2 is the aim of nocturnal non-invasive ventilation in stable COPD patients with chronic hypercapnia. PCO2 is normally measured non-invasively using a transcutaneous probe during overnight studies.
Percent of night time spent in hypercapnia | Overnight (about 8 hours)
  Hypercapnia is defined as PtcCO2 > 45 mm Hg. The aim of non-invasive ventilation in stable COPD patients is to reduce the time spent with PCO2 levels above the physiological range.

SECONDARY OUTCOMES:
Mean peripheral oxygen saturation (SpO2) | Through study completion, an average of 8 hours
  Peripheral oxygen saturation in a non-invasive measure of oxygenation, which is routinely evaluated in sleep and ventilation trials.
Desaturation | Through study completion, an average of 8 hours
  Desaturations are common complications in respiratory disorders. A desaturation is commonly defined by a reduction in SpO2 < 90%. The investigators computed the percent of night time in which SpO2 was < 90% and the Oxygen Desaturation Index (number of desaturations per hour).
Number of ineffective efforts per hour (IE) | Through study completion, an average of 8 hours
  Ineffective efforts are defined as inspiratory efforts that are not supported by the ventilator. They are indicative of patient-ventilator asynchrony, they may be associated with tidal expiratory flow limitation and they increase work of breathing and cause discomfort.
Sleep quality | Through study completion, an average of 8 hours
  Sleep quality is a key outcome during overnight studies. Nocturnal non-invasive ventilation may affect sleep quality in two ways: 1) it may improve it by reducing sleep-related respiratory problems; 2) it may worsen it if the ventilation mode causes discomfort to the patient. Sleep quality was evaluated by full laboratory polysomnography. Sleep stages were identified on epochs lasting 30 seconds by a trained operator blind to the study arms. Sleep quality was quantified using the following parameters: Sleep efficiency (percent of night time asleep), percentage of sleep time spent in phase 3 sleep and in REM sleep, number of awakenings per hour.
EPAP | Through study completion, an average of 8 hours
  The expiratory positive airway pressure (EPAP) is the parameter that is adjusted in the experimental arm. The ventilator automatically titrates EPAP to the minimum value able to abolish expiratory flow limitation.
Breathing pattern | Through study completion, an average of 8 hours
  Tidal volume, respiratory rate, minute ventilation, and inspiratory to expiratory time ratio are the breathing pattern parameters that the respiratory control system adjusts to achieve an adequate gas exchange while minimizing work of breathing. Non-invasive ventilation interacts with and supports breathing pattern.
Difference between mean inspiratory and expiatory reactance | Through study completion, an average of 8 hours
  The difference between mean inspiratory and expiatory reactance is measured using the forced oscillation technique. The difference between mean inspiratory and expiratory reactance is an index of tidal expiratory flow limitation. Values > 2.8 cmH2O*s/L are indicative of tidal expiratory flow limitation.
Mean inspiratory resistance | Through study completion, an average of 8 hours
  Mean inspiratory resistance is measured using the forced oscillation technique. Inspiratory resistance is an index of airway obstruction, which increases work of breathing and contributes to the development of flow limitation.
Mean inspiratory reactance | Through study completion, an average of 8 hours
  Mean inspiratory reactance is measured using the forced oscillation technique.
Sleep related respiratory event | Through study completion, an average of 8 hours
  During full laboratory polysomnography the respiratory activity is monitored and sleep related respiratory events are analysed, such as apneas, hypopnea, with a breakdown into central, peripheral or mixed events.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele L Dellacà, Prof., Principal Investigator — Politecnico di Milano
Locations (1):
- Divisione di Pneumologia, Fondazione S. Maugeri, IRCCS, Lumezzane, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milesi I, Porta R, Barbano L, Cacciatore S, Vitacca M, Dellaca RL. Automatic tailoring of the lowest PEEP to abolish tidal expiratory flow limitation in seated and supine COPD patients. Respir Med. 2019 Aug;155:13-18. doi: 10.1016/j.rmed.2019.06.022. Epub 2019 Jun 23. PMID 31276979
- [Derived] Zannin E, Milesi I, Porta R, Cacciatore S, Barbano L, Trentin R, Fanfulla F, Vitacca M, Dellaca RL. Effect of nocturnal EPAP titration to abolish tidal expiratory flow limitation in COPD patients with chronic hypercapnia: a randomized, cross-over pilot study. Respir Res. 2020 Nov 18;21(1):301. doi: 10.1186/s12931-020-01567-x. PMID 33208164